CLINICAL TRIAL: NCT05381935
Title: An Open-Label, Multicenter, First-in-Human, Dose Escalation and Expansion, Phase 1 Study of ES014 in Subjects With Locally Advanced or Metastatic Solid Tumors
Brief Title: A Study of ES014 (Anti-CD39/TGF-β Bispecific Antibody) in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor's clinical development strategy adjustment
Sponsor: Elpiscience Biopharma, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ES014-1001
Record Dates: First submitted 2022-05-11; First posted 2022-05-19 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 dose escalation (Experimental): ES014 doses will be escalated in patients with advanced solid tumors with approximately 30 subjects.
  Interventions: Drug: ES014
- Part 2 dose expansion (Experimental): Part 2 of the study will consist of 3 expansion cohorts for pancreatic ductal adenocarcinoma (Cohort 2A), NSCLC (Cohort 2B), and colorectal adenocarcinoma (Cohort 2C) with 10 subjects per expansion cohort respectively at the recommended optimal biological dose determined in Part 1 dose escalation.
  Interventions: Drug: ES014

INTERVENTIONS:
Drug: ES014 — ES014 is administered via intravenous infusion, once every 14 days, every 28 days as a treatment cycle for a maximum treatment duration per patient of 2 years.
  Arms: Part 1 dose escalation
Drug: ES014 — ES014 is administered via intravenous infusion, once every 14 days, every 28 days as a treatment cycle for a maximum treatment duration per patient of 2 years.
  Arms: Part 2 dose expansion

SUMMARY:
The purpose of this first-in-human, open-label, multicenter, non-randomized study designed to determine the maximum tolerated dose (MTD)/maximum administered dose (MAD), optimal biological dose (OBD), and recommended phase 2 dose (RP2D) of ES014 by evaluating the safety, tolerability, PK, pharmacodynamics, and preliminary clinical activity of ES014 administered intravenously to subjects with advanced solid tumors.

DETAILED DESCRIPTION:
Adenosine and transforming growth factor-β (TGF-β) are two key immune suppressors in the tumor microenvironment (TME) that cause broad immune suppression resulting in resistance to current checkpoint inhibitor immunotherapies. The bifunctional antibody-fusion protein ES014 was created by fusing the TGF-β receptor II ectodomain to an antibody targeting human ectonucleoside triphosphate diphosphohydrolase-1 (ENTPD1, CD39, UniprotKB: P49961). ES014 simultaneously neutralizes autocrine/paracrine TGF-β and inhibits the enzymatic activity of CD39, which results in the stabilization of pro-inflammatory extracellular adenosine triphosphate (eATP) and the restoration of anti-tumor immunity by impairing the accumulation of immune suppressive adenosine and TGF-β within the TME.

ELIGIBILITY:
Key Inclusion Criteria

1. To be eligible for study entry, subjects must satisfy all of the following criteria:
2. Capable of giving signed informed consent.
3. Part 1: Histological or cytological documentation of unresectable locally advanced or metastatic solid tumors, if 1) disease has progressed despite standard therapy, and no further standard therapy exists; or 2) standard therapy has proven to be ineffective or intolerable.

   Part 2: Histological or cytological documentation of PDAC (Cohort 2A), CRC (Cohort 2B), or NSCLC (Cohort 2C), with unresectable locally advanced or metastatic disease, if 1) disease has progressed despite standard therapy, and no further standard therapy exists; or 2) standard therapy has proven to be ineffective or intolerable.
4. Provide tumor tissue samples (minimum 10 unstained FFPE slides) obtained from the initial diagnosis to study entry.
5. At least one measurable lesion per RECIST v1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1.

   * Part 1: ECOG PS 0-1.
   * Part 2: ECOG PS 0-2.
7. Life expectancy of at least 12 weeks.
8. Adequate hematologic, hepatic, renal and coagulation functions per protocol
9. Male and female subjects of childbearing potential must be willing to completely abstain or agree to use a highly effective method of contraception

Key Exclusion Criteria

1. Any prior therapy targeting CD39, CD73, adenosine A2A receptor, or TGF-β.
2. Receipt of any investigational agents or devices within 4 weeks prior to the first dose of study drug.
3. Prior treatment with the following therapies:

   1. Anticancer therapy within 30 days or 5 half-lives of the drug prior to the first dose of study drug, whichever is shorter. At least 14 days must have elapsed between the last dose of prior anticancer agent and the first dose of study drug is administered. Exception: hormonal and/or hormonal replacement therapy.
   2. A wash out of at least 2 weeks before the start of study drug for radiation to the extremities and 4 weeks for radiation to the chest, brain, or visceral organs is required.
4. Prior allogeneic or autologous bone marrow transplantation or solid organ transplantation.
5. Toxicity from previous anticancer treatment per protocol.
6. Treatment with systemic immunosuppressive medications within 4 weeks prior to the first dose of study drug.
7. Subjects who received transfusion of blood products (including platelets or red blood cells), G-CSF, GM-CSF, recombinant erythropoietin, or recombinant thrombopoietin within 14 days prior to the first dose of study treatment.
8. Major surgery within 4 weeks prior to the first dose of study treatment.
9. Live vaccine therapies within 4 weeks prior to the first dose of study treatment.
10. Recent history of allergen desensitization therapy within 4 weeks prior to the first dose of study treatment.
11. Known allergies to CHO-produced antibodies, which in the opinion of the Investigator suggests an increased potential for an adverse hypersensitivity to ES014.
12. Invasive malignancy or history of invasive malignancy other than disease under study within the last two years per protocol.
13. CNS metastases.
14. Active autoimmune disease or documented history of autoimmune disease that required systemic steroids or other immunosuppressive medications per protocol.
15. Active interstitial lung disease (ILD) or pneumonitis or a history of ILD or pneumonitis requiring treatment with steroids or other immunosuppressive medications.
16. Active infection requiring systemic therapy, known human immunodeficiency virus (HIV) infection, or positive test for hepatitis B active infection (HBsAg) or hepatitis C active infection (hepatitis C antibody).
17. Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones, liver metastases, or otherwise stable chronic liver disease per investigator assessment).
18. History or evidence of cardiac abnormalities per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-21 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The frequency and severity of adverse events of ES014 | 1-3 years
  Adverse events will be assessed and assigned by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
  [Time Frame: 1-3 years]
Dose Limiting Toxicity of ES014 | Assessed during first 28 days of treatment
  Evaluation of dose-limiting toxicity (DLT)
Optimal biological dose (OBD) of ES014 | 1-3 years
  The OBD of ES014 will be determined

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) of ES014 | 1-3 years
  Maximum observed serum concentration (Cmax) of ES014 will be measured.
Trough observed serum concentration (Ctrough) of ES014 | 1-3 years
  Trough observed serum concentration (Ctrough)of ES014 will be measured.
Area under the serum concentration time curve (AUC) of ES014 | 1-3 years
  Area under the serum concentration time curve (AUC) of ES014 will be measured
Time to Cmax (Tmax) of ES014 | 1-3 years
  Time to Cmax (Tmax) of ES014 will be measured
The terminal elimination half life of ES014 | 1-3 years
  The terminal elimination half-life (t 1/2) of ES014 will be measured
The clearance of ES014 | 1-3 years
  A pharmacokinetic measurement of the volume of plasma from which ES014 is completely removed per unit time
The volume of distribution of ES014 | 1-3 years
  The amount of of ES014 in the body divided by the plasma concentration will be measured
The immunogenicity of ES014 | 1-3 years
  The presence and the frequency of anti-drug antibodies (ADA) against ES014 will be measured
The antitumor activity of ES014 | 1-3 years
  Tumor response will be measured by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1) by Investigator assessment

CONTACTS AND LOCATIONS:
Overall Officials: Elpiscience Biopharma, Ltd., Study Director — Elpiscience Biopharma, Ltd.

IPD SHARING:
Plan to Share IPD: No